CLINICAL TRIAL: NCT03147027
Title: Catheter Ablation for Nonsustained Ventricular Tachycardia in Patients With Ischemic Cardiomyopathy
Acronym: nsVT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Principal Investigator, Heinrich-Heine University, Duesseldorf
Other Study IDs: 15-007
Record Dates: First submitted 2017-05-05; First posted 2017-05-10 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Ventricular Tachycardia; Ischemic Cardiomyopathy; Reduced LVEF
Keywords: ischemic cardiomyopathy; prophylactic ablation
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Dosage Forms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VT ablation group
  Interventions: Procedure: VT ablation
- medication group
  Interventions: Other: medication

INTERVENTIONS:
Procedure: VT ablation — Substrate mapping for VT will be performed with the CARTO electroanatomical system.
  Groups: VT ablation group
Other: medication — medication to prevent sustained VT and ICD therapies
  Groups: medication group

SUMMARY:
Despite established implantable cardioverter-defibrillator (ICD) therapy and catheter ablation for sustained ventricular tachycardia (VT) in patients with ischemic heart disease (IHD) and reduced left ventricular ejection fraction (LVEF), the efficacy of catheter ablation in patients with nonsustained VT has been not yet clarified. The incidence of appropriate ICD therapy itself has been reported to be a worse prognostic factor in patients with reduced LVEF. Therefore theoretically the inhibition of these ventricular incidences can result in the prognostic improvement.To suppress ventricular arrhythmias aside from antiarrhythmic agents, catheter ablation has been developed prominently in this decade along with the technological improvement such as irrigated ablation catheters, three-dimensional mapping systems, multi-polar catheters, and image integration system with CT and MRI. The rationale of this trial is to study the efficacy of the eradication of arrhythmogenic substrate in ischemic cardiomyopathy with reduced LVEF and nonsustained VT on prevention of the occurrence of sustained VT/VF and ICD therapies.

ELIGIBILITY:
Inclusion Criteria:

* left ventricular ejection fraction (TTE or MRI) ≤40%
* diagnosed ischemic heart disease
* nonsustained monomorphic VT with more than 5 beats in the record of the implantable cardioverter-defibrillator or in any means of electrocardiogram (ECG) including ECG monitor and holter monitoring
* ICD implantation with primary preventive indication

Exclusion Criteria:

* ICD implantation within 2 months
* previously documented sustained VT/VF (over 30 seconds) or adequate ICD shock
* no written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with nonsustained VT and ischemic cardiomyopathy and reduced LVEF
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
occurrence of sustained VT/VF or ICD therapy | time from randomization to occurrence of any sustained VT/VF within 24 months
  occurrence of sustained VT/VF or ICD therapy including ATP and shock

SECONDARY OUTCOMES:
survival free from clinical events | time from randomization to 24 months
  survival free from clinical events (death, syncope, hospital admission due to cardiac problems, and VT storm, defined as more than three VT episodes in 24 hours)
number of appropriate ICD therapies | time from randomization to 24 months
  number of appropriate ICD therapies (ATP or shock)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany